CLINICAL TRIAL: NCT00785278
Title: Computationally Quantifying Wheelchair Set-Up to Minimize Peak Shoulder Joint Forces Throughout Manual Wheelchair Propulsion: A Pilot Study
Brief Title: Adjusting Wheelchair Set-Up to Minimize Shoulder Joint Forces During Propulsion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Responsible Party: Sarah R. Dubowsky, Ph.D., Postdoctoral Fellow, Kessler Medical Rehabilitation Research and Education Center
Other Study IDs: R-619-08
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2008-11-05 (Estimated); Status verified 2008-11

CONDITIONS: Paraplegia; Upper Limb Pain
Keywords: Wheelchair Set-Up; Shoulder Joint Forces; Manual Wheelchair Users; Paraplegia; Upper Limb Pain; Secondary Injury to Spinal Cord Injury; Biomechanics
MeSH Terms: conditions — Paraplegia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Able-bodied participants: Able-bodied individuals will be asked to propel a wheelchair at a self-selected speed for a period of time during which data will be collected on their propulsion biomechanics. It is assumed, for the purpose of the study, that un-learned able-bodied individuals learning to propel a wheelchair reflect newly injured individuals who are just getting accustomed to a new chair.
- 2: Participants with paraplegia: Individuals who are at least 1-year post injury and have used a manual wheelchair as their primary means of locomotion during this time, will be assumed to be, for the purpose of this study, experienced wheelchair users.

SUMMARY:
Individuals who use a manual wheelchair depend upon their upper limbs to provide a means of locomotion during completion of their activities of daily living. As a result of greater than normal usage of the upper limbs, shoulder pain and pathology is common among manual wheelchair users. Accordingly, proper wheelchair set-up may be paramount to preventing injuries and maintaining comfort during locomotion.

The purpose of this research study is to create a subject-specific computer model of wheelchair propulsion to provide information on wheelchair set-up (in particular, axle placement). The primary objective of this study is to investigate the effect of wheelchair set-up on shoulder joint forces during wheelchair propulsion; the secondary objective is to develop a predictive model to identify differences in shoulder joint forces that result from altering the axle position and seating set-up in user's wheelchairs.

The hypothesis of the study is that outputs from a patient-specific model will reveal that the current axle position for each subject results in peak shoulder joint forces that are greater than those predicted from an altered axle position (determined by the model). The overall goal is to then adjust each manual wheelchair user's axle placement to one that minimizes the magnitude of shoulder joint forces throughout propulsion. It is intended that in doing so, the repetitive strain injuries associated with manual wheelchair propulsion may be reduced, prolonging a pain-free way of life for this population.

ELIGIBILITY:
Experienced Wheelchair Users:

Inclusion Criteria:

* Have a neurological impairment secondary to a spinal cord injury which occurred over 1 year prior to the start of the study;
* SCI at or below T1 (complete or incomplete);
* Use a manual wheelchair as a primary means of mobility (at least 40 hrs. per week but not necessarily always in motion);
* SCI after age 18
* Have 24 inch diameter wheels with quick-release axles.

Exclusion Criteria:

* History of fractures or dislocations in the arms including the shoulder, elbow, and wrist;
* Upper limb dysthetic pain as a result of a syrinx or reflex sympathetic dystrophy;
* Pregnant women;
* Shoulder pain that a MWU describes as limiting their ability to propel a manual wheelchair;
* History of neurologic disorder other than spinal cord injury (e.g. brain injury).

Inexperienced Manual Wheelchair Users:

Inclusion Criteria:

* Be between the ages of 18 and 65 years of age.

Exclusion Criteria:

* History of fractures or dislocations in the arms including the shoulder, elbow, and wrist;
* Have a musculoskeletal disorder;
* Pregnant women;
* Shoulder pain that limits their ability to propel a manual wheelchair.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The racial, gender and ethnic characteristics of the proposed subject population reflects the demographics of Northern New Jersey and the surrounding area and/or the patient population of the Kessler Medical Rehabilitation Research and Education Center (KMRREC). Subjects will be recruited from database search and word of mouth.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-10 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Peak shoulder joint forces | During the propulsive phase of the push stroke at the time of data collection

SECONDARY OUTCOMES:
Propulsion Speed | Measured during the data collection process
Horizontal and Vertical Axle Placement | Measured prior to data collection on each test day

CONTACTS AND LOCATIONS:
Overall Officials: Sarah R. Dubowsky, Ph.D., Principal Investigator — Kessler Medical Rehabilitation Research and Education Center
Locations (1):
- Kessler Medical Rehabilitation Research and Education Center, West Orange, New Jersey, United States